CLINICAL TRIAL: NCT03176836
Title: Novel Approaches to Molecular and Clinical Surveillance in Li-Fraumeni Syndrome - Pilot Study.
Brief Title: Li-Fraumeni Syndrome Imaging Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrea Doria, Radiologist, Senior Scientist, Research Director, Department of Diagnostic Imaging, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000053416
Record Dates: First submitted 2017-05-11; First posted 2017-06-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Li-Fraumeni Syndrome
MeSH Terms: conditions — Li-Fraumeni Syndrome | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI Imaging (Experimental): Participants will be imaged with the standard MRI technique (STIR-MRI) and also new MRI techniques called "diffusion weighted" or "DW" MRI and Positron Emission Tomography (PET)-MRI. PET-MRI will be indicated if the results from the routine MRI and DW MRI are contradictory or if laboratory results do not correspond to the standard MRI and DW MRI results.
  Interventions: Diagnostic Test: Whole body STIR MRI; Diagnostic Test: DW-MRI; Diagnostic Test: PET-MRI

INTERVENTIONS:
Diagnostic Test: Whole body STIR MRI — Standard technique that detects abnormalities related to excess of water in tissues (edema).
Diagnostic Test: DW-MRI — MRI technique that analyzes areas of dead cells within tissues, present in some types of tumor.
Diagnostic Test: PET-MRI — MRI technique that detect's the cells' use of glucose, more intensely in harmful cells.

SUMMARY:
Li-Fraumeni Syndrome (LFS) is a cancer predisposition disorder in which most affected individuals develop cancer during their lifetime. The majority of LFS patients carry a mutation in a gene called TP53, whose normal function is to control cell growth and prevent cells with damaged DNA from becoming cancerous. There is currently no way to determine when, where or what type of tumour will develop. This project will use novel techniques utilizing magnetic resonance imaging (MRI) to determine how sensitive they are at detecting very small tumors and how specific they are in terms of distinguishing malignant tumors from benign tumors.

ELIGIBILITY:
Inclusion Criteria:

* LFS kindreds who either carry a known TP53 mutation or are obligate mutation carriers

Exclusion Criteria:

* General contraindications for an MRI scan (ferromagnetic prostheses, pacemaker, or other implants incompatible with the magnetic field of the MR scanner), claustrophobia.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of imaging traits on suspected tumors | Through study completion, an average of 2 years
  Imaging traits include: signal heterogeneity, mass effect, and neurovascular bundle involvement (recorded on STIR MRI); necrosis, and signal/necrosis ratio (recorded on STIR and DW MRI): FDG metabolic activity and uptake (PET-MRI) or other additional imaging findings. Results will be combined and analyzed for "extraction" of imaging-gene expression phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Doria, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No